CLINICAL TRIAL: NCT00601900
Title: Endocrine Therapy With or Without Anti-VEGF Therapy: A Randomized, Phase III Trial of Endocrine Therapy Alone or Endocrine Therapy Plus Bevacizumab (NSC 704865) for Women With Hormone Receptor-Positive Advanced Breast Cancer
Brief Title: Tamoxifen Citrate or Letrozole With or Without Bevacizumab in Treating Women With Stage IIIB or Stage IV Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00477; NCI-2009-00477 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB-40503; CDR0000584091; CALGB 40503/CTSU 40503; CALGB-40503 (Other: Alliance for Clinical Trials in Oncology); CALGB-40503 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2008-01-18; First posted 2008-01-28 (Estimated); Results first posted 2016-08-23 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Invasive Breast Carcinoma; Recurrent Breast Carcinoma; Stage III Breast Cancer AJCC v6; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Letrozole; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (endocrine therapy with monoclonal antibody) (Experimental): Patients receive endocrine therapy* (tamoxifen citrate* or letrozole) PO QD on days 1-21 and bevacizumab 15 mg/kg IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Other: Questionnaire Administration; Drug: Tamoxifen Citrate
- Arm II (endocrine therapy) (Active Comparator): Patients receive endocrine therapy* (tamoxifen citrate* or letrozole) PO QD on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Letrozole; Other: Questionnaire Administration; Drug: Tamoxifen Citrate

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm I (endocrine therapy with monoclonal antibody)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Letrozole — Given PO
  Other Names: CGS 20267; CGS-20267; CGS20267; Femara; Fempro
Other: Questionnaire Administration — Ancillary studies
Drug: Tamoxifen Citrate — Given PO
  Other Names: Apo-Tamox; Clonoxifen; Dignotamoxi; Ebefen; Emblon; Estroxyn; Fentamox; Gen-Tamoxifen; Genox; ICI 46,474; ICI 46474; ICI-46474; ICI46474; Jenoxifen; Kessar; Ledertam; Lesporene; Nolgen; Noltam; Nolvadex; Nolvadex-D; Nourytam; Novo-Tamoxifen; Novofen; Noxitem; Oestrifen; Oncotam; PMS-Tamoxifen; Soltamox; TAM; Tamax; Tamaxin; Tamifen; Tamizam; Tamofen; Tamoxasta; Tamoxifeni Citras; Zemide

SUMMARY:
This randomized phase III trial studies tamoxifen citrate or letrozole together with bevacizumab to see how well it works compared with tamoxifen citrate or letrozole alone in treating women with stage IIIB or stage IV breast cancer. Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen citrate or letrozole may fight breast cancer by blocking the use of estrogen by the tumor cells. Immunotherapy with monoclonal antibodies, such as bevacizumab, may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether giving hormone therapy is more effective with or without bevacizumab in treating advanced breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival of letrozole therapy alone with the combination of letrozole therapy plus bevacizumab as first-line treatment in women with estrogen- and/or progesterone-receptor-positive advanced breast cancer.

SECONDARY OBJECTIVES:

I. To compare the proportion of patients receiving letrozole alone, who remain progression-free at 6 and 12 months, to those receiving letrozole plus bevacizumab.

II. To compare the incidence of objective response (complete response [CR] + partial response [PR]) in patients receiving letrozole with and without bevacizumab, as determined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, excluding patients with non-measurable disease.

III. To compare the incidence of clinical benefit (CR + PR + stable disease >= 6 months) in patients receiving letrozole with and without bevacizumab.

IV. To compare the duration of objective response in patients receiving letrozole with and without bevacizumab.

V. To compare the time to treatment failure in patients receiving letrozole with and without bevacizumab.

VI. To compare the overall survival of patients receiving letrozole with and without bevacizumab, including the probability of survival until 36 months.

VII. To compare toxicity levels between the bevacizumab arm and the arm without bevacizumab in both the letrozole-treated patients and in the tamoxifen-treated patients.

VIII. To compare progression-free survival and overall survival of all patients receiving endocrine therapy with and without bevacizumab (by combining both letrozole and tamoxifen* patient subgroups).

CORRELATIVE OBJECTIVES:

I. To compare baseline and changes in serial levels of circulating endothelial cells and circulating tumor cells in patients treated with endocrine therapy alone or endocrine therapy plus bevacizumab, and to explore the relationship of these markers with progression free survival.

II. To conduct proteomic analysis of longitudinal samples from patients with advanced-stage disease undergoing hormonal therapy to define new serum-based biomarkers related to disease activity.

III. To identify biologic correlates that will predict progression-free survival (PFS) and response to therapy.

IV. To conduct pharmacogenomic assessment of candidate variants in the VEGF, CYP2D6, and CYP19 genes and evaluate their association with PFS and other study outcomes.

V. To identify single nucleotide polymorphisms (SNPs) associated with progression free survival in the genome-wide approach (GWAS).

VI. To identify factors other than chronological age that predict the risk of grade 3, 4 or 5 toxicity with bevacizumab and endocrine therapy by means of functional age assessment measures.

VII. To perform an exploratory analysis of the ability of the other factors included in the functional age assessment (either individual or in combination), to predict the risk of grade 3, 4 or 5 toxicity.

VIII. To evaluate longitudinal changes in the parameters of the factors described in objective VI while on therapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

NOTE: The placebo-controlled portion of the study was canceled on 5-15-10.

ARM I: Patients receive endocrine therapy* (tamoxifen citrate or letrozole) orally (PO) once daily (QD) on days 1-21 and bevacizumab intravenously (IV) over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive endocrine therapy* (tamoxifen citrate or letrozole) PO QD on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 6 months for the first 2 years and then annually for up to 3 years.

* NOTE: As of 5/15/2011, patients only receive letrozole.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of invasive cancer of the female breast in either the primary or metastatic setting

  * Stage IV disease or stage IIIB disease (using American Joint Committee on Cancer [AJCC] criteria, 6th edition) not amenable to local therapy
* Patients may not have a "currently active" second malignancy other than non-melanoma skin cancers; patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse
* Tumors (from either primary or metastatic sites) must express estrogen receptor (ER) and/or progesterone receptor (PgR) in >= 1% of cells will be considered positive
* Postmenopausal women are eligible for this trial; before study registration, menopausal status must be defined according to the criteria below:

  * Age >= 55 years and one year or more of amenorrhea
  * Age < 55 years and one year or more of amenorrhea, with an estradiol assay < 20 pg/ml
  * For women age < 55 with prior hysterectomy but intact ovaries, with an estradiol assay < 20 pg/ml
  * Surgical menopause with bilateral oophorectomy (at least 28 days must elapse from surgery to time of study registration)
  * Ovarian suppression on a luteinizing hormone-releasing hormone (LH-RH) agonist
* Premenopausal women who do not meet the postmenopausal criteria above are also eligible, but are required to undergo ovarian suppression; this can be initiated any time prior to or on day 1 of protocol therapy, regardless of chosen endocrine therapy, and will continue for the duration of protocol therapy
* Patients must have measurable or non-measurable disease by RECIST criteria, with radiologic scans within 28 days of study registration

  * Measurable disease: lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 2.0 cm with conventional techniques or as >= 1.0 cm with spiral computed tomography (CT) scan
  * Non-measurable disease: all other lesions, including small lesions (longest diameter < 2.0 cm with conventional techniques or < 1.0 cm with spiral CT scan) and truly non-measurable lesions
  * Lesions that are considered non-measurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Prior endocrine therapy is not required

  * Prior endocrine therapy in the metastatic setting is not permitted (unless tamoxifen or an aromatase inhibitor was initiated within 4 weeks prior to registration to facilitate enrollment of patients who recently started first-line endocrine therapy for metastatic breast cancer); if prior letrozole therapy was initiated within the past 4 weeks, the patients should remain on letrozole as the study therapy; patients who began therapy with tamoxifen, anastrozole or exemestane must switch to letrozole to be eligible to participate in this study
  * Prior endocrine therapy in the adjuvant setting is permitted; there is no time restriction for how long the patient must be on the adjuvant endocrine therapy, nor is there a time restriction for how long the patient needs to be off prior adjuvant endocrine therapy before beginning protocol therapy on 40503
  * Prior treatment with ovarian suppression is allowed in either the adjuvant or metastatic setting; if medical ovarian suppression is being administered it can be initiated any time prior to or at the start of protocol therapy, and continued throughout the duration of the trial; surgical castration with bilateral oophorectomy must be performed at least 28 days prior to study registration (due to concerns of poor wound healing on bevacizumab)
* Patients may not have received any prior anti-VEGF or VEGFR tyrosine kinase inhibitor therapy
* Prior radiotherapy must have been completed and all toxicities resolved at least two weeks prior to registration
* Chemotherapy in the adjuvant or neoadjuvant setting is permitted; at least twelve months prior to registration must have elapsed since the completion of adjuvant or neoadjuvant chemotherapy and all toxicities must have resolved; taxane-related neurotoxicity must have resolved to sensory grade < 2 and no motor neuropathy of any grade is allowed
* Patients may have received one prior chemotherapy regimen for metastatic disease; the final dose of prior chemotherapy must have been administered at least 3 weeks prior to study registration
* Treatment with bisphosphonates is allowed and recommended as per American Society of Clinical Oncology (ASCO) guidelines
* Patients must not have had a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study registration, and must have fully recovered from any such procedure
* Patients must not have anticipation of need for major surgical procedure during the course of the study
* Patients must not have had a core biopsy or other minor surgical procedure, within 7 days prior to study registration; placement of a vascular access device is allowed within 7 days of registration
* Patients must not have a history of abdominal fistula, or intra-abdominal abscess within 6 months prior to study registration
* Patients with a history of gastrointestinal (GI) perforation within 12 months prior to registration are not eligible
* Patients with a history of significant bleeding episodes (e.g., hemoptysis, upper or lower GI bleeding) within 6 months prior to registration are not eligible
* Patients must not have clinically significant cardiovascular disease that includes the following:

  * Uncontrolled hypertension defined as systolic blood pressure > 150 and/or diastolic blood pressure > 90 mmHg on antihypertensive medications or any prior history of hypertensive crisis or hypertensive encephalopathy
  * History of myocardial infarction or unstable angina within past 6 months
  * New York Heart Association (NYHA) grade 2 or greater congestive heart failure
  * Symptomatic peripheral vascular disease
  * Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or arterial thrombotic events
* Full dose anticoagulation therapy is allowed for the treatment of prior conditions such as venous thrombosis or atrial fibrillation, but not for the treatment of prior arterial thrombotic events; patients on full dose anticoagulants must be on a stable dose of warfarin and have an in-range international normalized ratio (INR) (usually between 2 and 3) or be on a stable dose of low-molecular weight (LMW) heparin; patients receiving antiplatelet agents are eligible, as are patients on daily prophylactic aspirin or anticoagulation for atrial fibrillation
* Patients may not have a history of stroke or transient ischemic attack within 6 months prior to study registration
* Patients with a history of seizures must be well controlled with standard medication
* Patients must not have known central nervous system (CNS) metastases or leptomeningeal disease (screening with brain imaging is not required for asymptomatic patients)
* In aromatase inhibitor (AI)-treated patients: no known allergies to imidazole drugs, (e.g. clotrimazole, ketoconazole, miconazole, econazole, sulconazole, tioconazole, or terconazole) or compounds structurally similar to bevacizumab
* In tamoxifen treated patients: no known allergies to selective estrogen receptor modulators (e.g. tamoxifen, raloxifene or toremifene) or compounds structurally similar to bevacizumab; for patients enrolled after Update #5, endocrine therapy will consist of letrozole only and this criterion will no longer apply
* Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status =< 1
* No serious, non-healing wound, ulcer, or bone fracture
* Life expectancy of >= 12 weeks
* All patients who are premenopausal (if not already receiving ovarian suppression therapy/surgical oophorectomy) must have a negative beta-human chorionic gonadotropin (beta-Hcg) prior to starting on study treatment; patients may not be pregnant or nursing at any time during the study; ovarian suppression is required in women of childbearing potential by the start of protocol therapy, and will continue for the duration of protocol therapy
* Granulocytes >= 1,000/ul
* Platelet count >= 100,000/ul
* Creatinine =< 2.0 mg/dL
* Bilirubin =< 1.5 times upper limit of normal (ULN) unless due to Gilbert's syndrome
* Transaminases (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) =< 2.5 times ULN
* International normalized ratio (INR) =< 1.6, unless on full dose warfarin
* Beta-Hcg negative in premenopausal women
* Urine protein =< 1+ or urine to plasma creatinine (UPC) < 1

  * Patients discovered to have >= 2+ proteinuria at baseline must undergo a 24-hour urine collection that must demonstrate < 1 g of protein/24 hr, or UPC ratio < 1 to allow participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2008-09-24 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2025-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S Rugo, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (522):
- United States (521):
  - Providence Hospital, Mobile, Alabama
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - East Bay Medical Oncology Hematology Medical Associates-Antioch, Antioch, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Adventist Health Cancer Care Center Chico, Chico, California
  - Community Cancer Institute, Clovis, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Marin General Hospital, Greenbrae, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - East Bay Medical Oncology Hematology Medical Associates Inc-Pleasant Hill, Pleasant Hill, California
  - John Muir Health Cancer Medical Group, Pleasant Hill, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - East Bay Medical Oncology Hematology Associates Inc, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Saint Helena Hospital, St. Helena, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists-Gainesville Cancer Center, Gainesville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Dublin Hematology Oncology Care PC, Dublin, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Eisenhower Army Medical Center, Fort Eisenhower, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Freeport Memorial Hospital/Leonard C Ferguson Cancer Center, Freeport, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Our Lady Bellefonte Hospital, Ashland, Kentucky
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Veterans Administration Medical Center-Baltimore, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Meritus Medical Center, Hagerstown, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente Lutherville - Timonium Medical Center, Lutherville, Maryland
  - Kaiser Permanente - Shady Grove Medical Center, Rockville, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Hospital, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Queens Hospital Center, Jamaica, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Highland Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island Inc, Cranston, Rhode Island
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Kaiser Permanente - Fair Oaks Medical Center, Fairfax, Virginia
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Providence Holy Family Hospital, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Cancer Care-Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Quintanilha JCF, Wang J, Sibley AB, Jiang C, Etheridge AS, Shen F, Jiang G, Mulkey F, Patel JN, Hertz DL, Dees EC, McLeod HL, Bertagnolli M, Rugo H, Kindler HL, Kelly WK, Ratain MJ, Kroetz DL, Owzar K, Schneider BP, Lin D, Innocenti F. Bevacizumab-induced hypertension and proteinuria: a genome-wide study of more than 1000 patients. Br J Cancer. 2022 Feb;126(2):265-274. doi: 10.1038/s41416-021-01557-w. Epub 2021 Oct 6. PMID 34616010
- [Derived] Martin M, Loibl S, Hyslop T, De la Haba-Rodriguez J, Aktas B, Cirrincione CT, Mehta K, Barry WT, Morales S, Carey LA, Garcia-Saenz JA, Partridge A, Martinez-Janez N, Hahn O, Winer E, Guerrero-Zotano A, Hudis C, Casas M, Rodriguez-Martin C, Furlanetto J, Carrasco E, Dickler MN; GEICAM Spanish Breast Cancer Group; GBG (German Breast Group); Alliance for Clinical Trials in Oncology (Alliance). Evaluating the addition of bevacizumab to endocrine therapy as first-line treatment for hormone receptor-positive metastatic breast cancer: a pooled analysis from the LEA (GEICAM/2006-11_GBG51) and CALGB 40503 (Alliance) trials. Eur J Cancer. 2019 Aug;117:91-98. doi: 10.1016/j.ejca.2019.06.002. Epub 2019 Jul 2. PMID 31276981
- [Derived] Li D, McCall LM, Hahn OM, Hudis CA, Cohen HJ, Muss HB, Jatoi A, Lafky JM, Ballman KV, Winer EP, Tripathy D, Schneider B, Barry W, Dickler MN, Hurria A. Identification of risk factors for toxicity in patients with hormone receptor-positive advanced breast cancer treated with bevacizumab plus letrozole: a CALGB 40503 (alliance) correlative study. Breast Cancer Res Treat. 2018 Sep;171(2):325-334. doi: 10.1007/s10549-018-4828-5. Epub 2018 May 22. PMID 29789969
- [Derived] Dickler MN, Barry WT, Cirrincione CT, Ellis MJ, Moynahan ME, Innocenti F, Hurria A, Rugo HS, Lake DE, Hahn O, Schneider BP, Tripathy D, Carey LA, Winer EP, Hudis CA. Phase III Trial Evaluating Letrozole As First-Line Endocrine Therapy With or Without Bevacizumab for the Treatment of Postmenopausal Women With Hormone Receptor-Positive Advanced-Stage Breast Cancer: CALGB 40503 (Alliance). J Clin Oncol. 2016 Aug 1;34(22):2602-9. doi: 10.1200/JCO.2015.66.1595. Epub 2016 May 2. PMID 27138575
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Endocrine Therapy With Monoclonal Antibody) | Arm II (Endocrine Therapy)
Started | 195 | 199
Completed | 195 | 196
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Endocrine Therapy With Monoclonal Antibody) | Arm II (Endocrine Therapy) | Total
Number analyzed (Participants) | 195 | 196 | 391
Age, Continuous [Median (Full Range); unit: years] | 55.5 [24.7 to 85.3] | 58.9 [29.0 to 87] | 57.7 [24.7 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 196 | 391
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 195 | 196 | 391
Endocrine Therapy Elected [Number; unit: participants]
  Letrozole | 174 | 174 | 348
  Tamoxifen | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The Primary Endpoint for this study was to compare the progression-free survival of letrozole therapy alone with the combination of letrozole therapy plus bevacizumab as first-line treatment in women with estrogen- and/or progesterone-receptor-positive advanced breast cancer. Progression-free survival (PFS) was defined as the time from randomization until disease progression or death, whichever occurs first. The median PFS was estimated using the Kaplan-Meier method. Progression was assessed per RECIST criteria, and defined as at least a 20% increase in the sum of the longest diameters of target lesions from baseline or the appearance of new lesions.
Time Frame: From randomization until disease progression or death whichever occurs first, assessed up to 5 years
Population: Per protocol, the analysis of the primary endpoint was restricted to patients that elected letrozole as endocrine therapy. Of the 348 patients electing Letrozole, 5 did not receive treatment (1 on Arm I, and 4 on Arm II). This left 343 patients (173 on the Arm I and 170 on Arm II) evaluable for the primary endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Endocrine Therapy With Monoclonal Antibody) | Arm II (Endocrine Therapy)
Number analyzed (Participants) | 173 | 170
months | 20.2 [17 to 24] | 15.6 [12.9 to 19.7]

2. Secondary Outcome: 12 Month Progression Free Survival Rate
Description: The 12 month progression-free survival rate was defined as the proportion of patients who were alive progression-free 12 months after registration into the study.
Time Frame: At 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Endocrine Therapy With Monoclonal Antibody) | Arm II (Endocrine Therapy)
Number analyzed (Participants) | 173 | 170
percentage of participants | 73 [66 to 80] | 61 [54 to 68]

3. Secondary Outcome: 6 Month Progression-Free Survival Rate
Description: The 6 month progression-free survival rate was defined as the proportion of patients who were alive progression-free 6 months after registration into the study.
Time Frame: At 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Endocrine Therapy With Monoclonal Antibody) | Arm II (Endocrine Therapy)
Number analyzed (Participants) | 173 | 170
percentage of participants | 87 [82 to 93] | 77 [71 to 83]

4. Secondary Outcome: Objective Response Rate
Description: Response was defined using RECIST criteria: Complete Response (CR): disappearance of all target lesions; Partial Response (PR) 30% decrease in sum of longest diameter of target lesions.
Time Frame: Assessed up to 5 years
Population: Per protocol, the analysis of this endpoint was restricted to patients that elected letrozole as endocrine therapy and began treatment with measureable disease. A total of 213 patients (Arm A:106; Arm B:107) had measureable disease. Of the 213, 197 (Arm A:98, Arm B:99) patients were assessed for response during treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Endocrine Therapy With Monoclonal Antibody) | Arm II (Endocrine Therapy)
Number analyzed (Participants) | 98 | 99
percentage of participants
  Complete Response (CR) | 4 | 7
  Partial Response (PR) | 65 | 42
  Stable Disease (SD) | 22 | 34

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from study entry to death from any cause. The median OS was estimated using the Kaplan-Meier method.
Time Frame: Assessed up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Endocrine Therapy With Monoclonal Antibody) | Arm II (Endocrine Therapy)
Number analyzed (Participants) | 173 | 170
months | 47.2 [39 to 56.8] | 43.9 [37.6 to 49.6]

6. Secondary Outcome: Duration of Tumor Response
Description: Defined by RECIST criteria.
Time Frame: From the time measurement criteria are met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 5 years
Reporting Status: Not Posted

7. Secondary Outcome: Probability of Surviving Until 36 Months
Time Frame: At 36 months
Reporting Status: Not Posted

8. Secondary Outcome: Site of Progression
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Secondary Outcome: Time-to-treatment Failure
Description: From randomization until first disease progression, early termination of protocol therapy due to toxicity or withdrawn consent, or going onto non-protocol therapy. Defined by RECIST criteria. The proportional hazards model will be used to compare the arms on time-to-treatment-failure
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Secondary Outcome: Treatment Related Toxicity
Description: Graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Tabulated by type, grade, and arm.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All patients that received study treatment and were analyzed for adverse events are included in this summary.
Arm/Group | Arm I (Endocrine Therapy With Monoclonal Antibody) | Arm II (Endocrine Therapy)
Serious Adverse Events (participants affected / at risk) | 56/195 | 30/196
Other Adverse Events (participants affected / at risk) | 174/195 | 145/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Endocrine Therapy With Monoclonal Antibody) (N=195) | Arm II (Endocrine Therapy) (N=196)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (8) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 3 (3)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1)
Fever (General disorders) | 6 (6) | 2 (2)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 2 (2)
Endocarditis infective (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 3 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intraoperative reproductive tract injury - Uterus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Small intestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Cardiac troponin T increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (31) | 12 (18)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 13 (15) | 4 (5)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (2)
Proteinuria (Renal and urinary disorders) | 18 (21) | 2 (3)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 20 (23) | 6 (6)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Endocrine Therapy With Monoclonal Antibody) (N=195) | Arm II (Endocrine Therapy) (N=196)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (12) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (16) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (2)
Left ventricular failure (Cardiac disorders) | 4 (4) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 2 (4)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 2 (4)
Dry eye syndrome (Eye disorders) | 1 (17) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (6) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 2 (5) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (29) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (20) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mouth necrosis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (19) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 2 (5) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (3) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 3 (5) | 0 (0)
Fatigue (General disorders) | 19 (69) | 12 (21)
Fever (General disorders) | 24 (32) | 15 (18)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (15) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 13 (27) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 2 (3)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis infective (Infections and infestations) | 0 (0) | 1 (2)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Gingival infection (Infections and infestations) | 1 (2) | 1 (1)
Infection (Infections and infestations) | 3 (3) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (4) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 7 (25) | 3 (4)
Skin infection (Infections and infestations) | 2 (3) | 1 (1)
Tooth infection (Infections and infestations) | 4 (6) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 10 (14) | 5 (11)
Ureteritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 10 (16) | 4 (5)
Vaginal infection (Infections and infestations) | 1 (1) | 2 (4)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (6) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 6 (8) | 1 (2)
Alanine aminotransferase increased (Investigations) | 4 (8) | 2 (6)
Alkaline phosphatase increased (Investigations) | 4 (9) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (14) | 3 (5)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 3 (7) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (3) | 0 (0)
INR increased (Investigations) | 2 (10) | 0 (0)
Leukocyte count decreased (Investigations) | 1 (12) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (14) | 1 (1)
Platelet count decreased (Investigations) | 3 (28) | 0 (0)
Weight loss (Investigations) | 5 (39) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (22) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (26) | 4 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Serum potassium increased (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (8) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 137 (1597) | 115 (1120)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (37) | 7 (23)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (16) | 2 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (14) | 6 (19)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 3 (6)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (12) | 2 (15)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Acoustic nerve disorder NOS (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5) | 2 (2)
Headache (Nervous system disorders) | 85 (409) | 58 (245)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 3 (7) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 2 (5)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (6) | 3 (4)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 5 (24) | 2 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 93 (818) | 13 (42)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 1 (6)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (16) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 (160) | 2 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (7) | 0 (0)
Hemorrhage (Vascular disorders) | 3 (4) | 0 (0)
Hot flashes (Vascular disorders) | 12 (46) | 8 (34)
Hypertension (Vascular disorders) | 115 (1029) | 61 (528)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 6 (7) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less